CLINICAL TRIAL: NCT06109376
Title: Efficacy and Safety of Endovascular Thrombectomy With Versus Without Hypothermia in Acute Large Vessel Occlusion Stroke: a Randomized Controlled Trial
Brief Title: Role of Hypothermia in Endovascular Stroke Thrombectomy
Acronym: COOLING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Xiangtan Central Hospital (Other)
Responsible Party: Principal Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COOLING
Record Dates: First submitted 2023-10-22; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Acute Ischemic
Keywords: endovascular thrombectomy; hypothermia; large vessel occlusion; randomized controlled trial
MeSH Terms: conditions — Ischemic Stroke; Hypothermia | interventions — Thrombectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermia (Experimental): Patients in Hypothermia group received hypothermia combined with endovascular thrombectomy.
  Interventions: Procedure: hypothermia; Procedure: thrombectomy
- Control (Active Comparator): Patients in Control group received endovascular thrombectomy alone.
  Interventions: Procedure: thrombectomy

INTERVENTIONS:
Procedure: hypothermia — In this trial, intra-arterial select cooling infusion is used to reduce brain tissue temperature to 33-35°C.
  Arms: Hypothermia
Procedure: thrombectomy — Thrombectomy includes treatment with stent retrievers and/or thromboaspiration, balloon angioplasty, stenting, intra-arterial thrombolysis, or the various combinations of these approaches.

SUMMARY:
Reducing or suspending the increase of the infarcted core, i.e., "freezing" the ischemic penumbra, may help improve the efficacy of mechanical thrombectomy. Hypothermia effectively reduces the metabolic level of brain tissue, may prolong the time window for recanalization therapy, and its multi-target therapeutic effect make it one of the most promising neuro-protection approach.

In recent years, hypothermia has been increasingly used to treat acute ischemic stroke. However, its role in acute ischemic stroke is unclear.

The objective of this trial is to investigate whether hypothermia combined with endovascular thrombectomy could add additional benefit without increasing the risk of adverse events such as pneumonia, intracerebral hemorrhage, and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years or more;
2. acute ischemic stroke within 24 hours from onset to randomization;
3. NIHSS ≥6 points before randomization;
4. Internal carotid artery, or the middle cerebral artery M1 or M2 occlusion confirmed by CTA/MRA/DSA;
5. Baseline ASPECTS score ≥ 3 and ≤8, or cerebral infarction core volume < 100ml;
6. The patient decides to undergo endovascular therapy;
7. The patient or patient's representative signs a written informed consent form.

Exclusion Criteria:

1. CT or MR evidence of hemorrhage;
2. Currently pregnant or lactating (women patients);
3. Allergy to radiographic contrast agents, or nitinol devices;
4. Arterial tortuosity and/or other arterial disease that would prevent the device from reaching the target vessel;
5. Multiple vessel occlusion (e.g., bilateral anterior circulation, or occlusion of both anterior and posterior circulation);
6. Preexisting neurological or psychiatric disease that would confound the neurological functional evaluations;
7. Previous bleeding disorders, severe heart, liver or kidney disease, or sepsis;
8. Brain tumors with mass effect (except meningiomas) that are radiographically pleasant;
9. Intracranial aneurysm, arteriovenous malformation;
10. Any terminal illness with life expectancy less than 6 months;
11. Participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale score (mRS) | 90 days post-randomization
  Modified Rankin scale score (mRS): scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death

SECONDARY OUTCOMES:
Excellent outcome | 90 days post-randomization
  Score of 0-1 on the modified Rankin scale
Functional independence | 90 days post-randomization
  Score of 0-2 on the modified Rankin scale
Moderate outcome | 90 days post-randomization
  Score of 0-3 on the modified Rankin scale
Early neurological improvement | 72 hours post-randomization
  Compared with baseline NIHSS, the 72h NIHSS score is reduced by 8 points or more, or the 72h NIHSS is 0~1 point
EQ-5D-5L scale score | 90 days post-randomization
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Successful reperfusion at final angiogram | At the end of angiography or procedure
  Successful reperfusion was defined as grade 2b to 3 on the extended Thrombectomy in the Cerebral Ischemia system.
Difference between baseline and within 48h after procedure of infarction core volume (ml) | 48 hours post-randomization
Reperfusion on follow-up CT or MR angiography | 48 hours post-randomization
Incidence of symptomatic intracranial hemorrhage (SICH) | 48 hours post-randomization
  using Heidelberg criteria to assess SICH
incidence of any intracranial hemorrhage (any ICH) | 48 hours post-randomization
90-day mortality | 90 days post-randomization
Difference of hematocrit between baseline and 24-hour post-randomization | 24-hour post-randomization
Non-hemorrhagic serious adverse event rate | 90 days post-randomization
  including pneumonia, respiratory failure, circulatory failure, cerebral herniation, secondary epilepsy, sepsis, renal failure, acute coronary syndrome, venous thrombosis, etc.
Complications related to operation and device | 90 days post-randomization
  vasospasm, arterial rupture, arterial dissection, vascular puncture point complications, etc.
Other serious adverse events | 90 days post-randomization

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, and Analytic Code will be shared after approval of a proposal from principal investigator 3 years after the trial results are revealed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after the trial results are revealed.
Access Criteria: after approval of a proposal from principal investigator